CLINICAL TRIAL: NCT00996268
Title: An Open-label Single Dose Randomized, Parallel Group Study Followed by Single-blind Repeat Dosing, to Compare the Relative Bioavailability of GSK2212836
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 113412
Record Dates: First submitted 2009-10-15; First posted 2009-10-16 (Estimated); Last update posted 2017-06-22 (Actual); Status verified 2017-06

CONDITIONS: Cardiovascular Disease
Keywords: hypertriglyceridemia; GSK2212836; relative bioavailability
MeSH Terms: conditions — Cardiovascular Diseases; Hypertriglyceridemia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Part A (Experimental): Three groups of sixteen healthy subjects will be randomized to single doses of 3 different formulations of GSK2212836.
  Interventions: Drug: GSK2212836
- Part B (Experimental): Four cohorts of at least 10 subjects will participate in a 2-week repeat dose period with 4 dose levels (based on data obtained in Part A) of the GSK2212836 test formulations or placebo.
  Interventions: Drug: GSK2212836

INTERVENTIONS:
Drug: GSK2212836 — Treatment A - GSK2212836 test formulation 1, Treatment B - GSK2212836 test formulation 2, or Treatment C -GSK2212836 marketed formulation.
  Arms: Part A
Drug: GSK2212836 — Treatment D - low dose of GSK2212836 test formulation, Treatment E - medium dose of GSK2212836 test formulation, Treatment F - high dose of GSK2212836 test formulation, Treatment G - GSK2212836 marketed formulation, or Placebo.
  Arms: Part B

SUMMARY:
Sixteen healthy subjects will be randomized to each of the 3 parallel treatment groups. Eligible subjects will check in to the clinical unit on Day -2 and have 24-hr pharmacokinetic collections on Day -1 and on Day 1. Once the pharmacokinetic parameters of the formulations have been analyzed, doses of GSK2212836 will be selected for further study in Part B. Subjects from Part A will participate in Part B.

Part B is a single blind, randomized, placebo controlled study that will consist of a 2-week repeat dose period with 3 dose levels and one dose of the marketed formulation of GSK2212836. Subjects will check in to the clinical unit on Day -3; will participate in a test meal on Day -2 and have 24-hr baseline pharmacokinetic profiles on Day -1 and Day 1. Subjects will be released from the clinic on Day 2, and return for daily dosing on Days 3 through 12. On Day 6, they will also have a brief outpatient visit. Subjects will check into the clinic again on the evening of Day 12, and on Day 13 they will again have 24-hr pharmacokinetic profiles collected. Subjects will be released from the clinical research unit on Day 14, following a test meal, triglyceride sampling and check-out assessments, and will be released from the study 5-10 days later after completing a follow up visit.

ELIGIBILITY:
Inclusion Criteria:

* AST, ALT, alkaline phosphatase and bilirubin less than 1.5xULN (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%).
* Healthy as determined by a responsible and experienced physician, based on a medical evaluation including [medical history, physical examination, laboratory tests and ECGs. A subject with a clinical abnormality or laboratory parameters outside the reference range for the population being studied may be included only if the Investigator and the GSK Medical Monitor agree that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures.
* Male or female between 18 and 50 years of age inclusive, at the time of signing the informed consent.
* A female subject is eligible to participate if she is of Child-bearing potential and agrees to use one of the contraception methods listed in the protocol.
* Body weight greater than or equal to 50kg (110 lbs) for men and greater than or equal to 45 kg for women and BMI within the range 24-34kg/m2 (inclusive).
* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.
* Average QTcB or QTcF < 450 msec; or QTc < 480 msec in subjects with Bundle Branch Block.

Exclusion Criteria:

* A positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result within 3 months of screening
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* A positive pre-study drug/alcohol screen.
* A positive test for HIV antibody.
* History of regular alcohol consumption within 6 months of the study defined as:
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* Exposure to more than four new chemical entities within 12 months prior to the first dosing day.
* Use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements (including St John's Wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of study medication, unless in the opinion of the Investigator and GSK Medical Monitor the medication will not interfere with the study procedures or compromise subject safety.
* Use of omega-3 fatty acid supplements and/or fish or fish oil products from screening until final assessment and unwilling to abstain from eating oily fish (salmon, albacore tuna, mackerel, sardines, etc.) during the course of the study.
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or GSK Medical Monitor, contraindicates their participation.
* History of sensitivity or known allergy to fish and /or shellfish.
* Where participation in the study would result in donation of blood or blood products in excess of 500 mL within a 56 day period.
* Pregnant females as determined by positive hCG test at screening (serum) or prior to dosing (urine).
* Lactating females.
* Unwillingness or inability to follow the procedures outlined in the protocol.
* Subject is mentally or legally incapacitated.
* History of sensitivity to heparin or heparin-induced thrombocytopenia.
* Unable to abstain from smoking tobacco- or use of nicotine-containing products while in the clinic.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 46 (Actual)
Dates: Start 2009-10-15 (Actual); Primary Completion 2010-01-04 (Actual); Study Completion 2010-01-04 (Actual)

PRIMARY OUTCOMES:
Part A: To determine the total (AUC(0 to infinity)) and peak (Cmax) exposure of GSK2212836 | 24 hours
Part B: PK parameters AUC(0-24h) and Cmax following 14 days of dosing with GSK2212836 | 14 days
Part A: To assess the relative bioavailability of GSK2212836 test capsules vs the reference formulation GSK2213836 | 24 hours
Part B: To estimate the accumulation and dose proportionality of GSK2212836 after repeat dosing of the test formulation | 14 days

SECONDARY OUTCOMES:
Part A: Safety and tolerability parameters following single doses of GSK2212836 test formulation including adverse events, clinical laboratory, ECGs and vital signs assessments. | 24 hours
Part A: Secondary PK parameters including: tmax, t1/2 and baseline-corrected AUC(0-24h) | 24 hours
Part B: Safety and tolerability parameters following repeat doses of GSK2212836 test formulation including adverse events, clinical laboratory, ECGs and vital signs assessments | 14 days
Part B: Secondary PK parameters including: tmax, t1/2 | 14 days

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Buffalo, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Hussey EK, Portelli S, Fossler MJ, Gao F, Harris WS, Blum RA, Lates CD, Gould E, Abu-Baker O, Johnson S, Reddy KK. Relative Bioavailability of an Emulsion Formulation for Omega-3-Acid Ethyl Esters Compared to the Commercially Available Formulation: A Randomized, Parallel-Group, Single-Dose Study Followed by Repeat Dosing in Healthy Volunteers. Clin Pharmacol Drug Dev. 2012 Jan;1(1):14-23. doi: 10.1177/2160763X11431107. PMID 27206142
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- See also: Results for study 113412 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/113412?search=study&study_ids=113412#rs
- Available data/document: Individual Participant Data Set: 113412 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 113412 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 113412 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 113412 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 113412 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 113412 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 113412 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register